CLINICAL TRIAL: NCT02731612
Title: A 6-Week Randomised, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy of Lurasidone Adjunctive Therapy in Improving Cognitive Functioning in Euthymic Bipolar Disorder Patients (ELICE-BD)
Brief Title: Study of the Efficacy of Lurasidone in Cognitive Functioning in Bipolar Patients
Acronym: ELICE_BD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lakshmi N Yatham (Other)
Responsible Party: Sponsor-Investigator, Lakshmi N Yatham, Prinicipal Investigator, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H16-00129
Record Dates: First submitted 2016-03-23; First posted 2016-04-07 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Cognition; Euthymic; Lurasidone
MeSH Terms: conditions — Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lurasidone (Experimental): Lurasidone 20 - 80 mg / day added to current treatment for 6 weeks.
  Interventions: Drug: lurasidone
- Placebo (Placebo Comparator): Placebo added to current treatment for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: lurasidone — Atypical Antipsychotic
  Other Names: Latuda
  Arms: Lurasidone
Other: Placebo — Inactive substance
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicentre, parallel-group study to assess the cognitive effects of lurasidone in bipolar I and II patients (manic depression) who are in remission from an episode. Participants who show cognitive impairment at the screening visit will be enrolled into the study and randomized at the baseline visit to receive either lurasidone or placebo adjunctive therapy in a 1:1 ratio for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 19 to 65 years inclusive.
2. Diagnostic and Statistical Manual of Mental Disorder, 5th Edition (DSM.5) diagnosis of Bipolar Type I or Type II Disorder, with or without a history of psychosis. BP II patients must have had 2 definite periods of hypomania in the last 5 years.
3. All patients must be taking either a mood stabilizer (i.e. lithium or valproate) (lamotrigine as a mood stabilizer is acceptable for bipolar 2 disorder patients only and not for bipolar I disorder) or an atypical antipsychotic or a combination of these (two mood stabilizers or a mood stabilizer plus an atypical antipsychotic), at therapeutic doses, for mood stabilization. Those taking two atypical antipsychotics are excluded. Combinations of these medications as outlined above, or the combination of any of them with lamotrigine 100-400 mg daily, or the combination of a mood stabilizer plus asenapine 5-20 mg/day, are also permitted.
4. All concomitant medication must be at a stable dose for two weeks prior to the randomization visit.
5. Clinically stable during the last 4 weeks as assessed by clinical interview.
6. A Montgomery Asberg Depression Rating Scale(MADRS) and Young Mania Rating Scale (YMRS) score less than or equal to 8.
7. Patients who show cognitive impairments (-0.50 SD or below) on either the Wechsler Adult Intelligence Scale-IV (WAIS-IV) -Coding subtest, or the Rey Auditory Verbal Learning Test (RAVLT) total learning score on trials 1 to 5 or immediate recall, at screening visit.
8. A WAIS-IV vocabulary scaled score >5 (equivalent to estimated IQ 80 or greater).
9. A sufficient level of the English or Japanese language.
10. Females who are postmenopausal for at least 1 year before the screening visit (confirmed by an FSH test) or are surgically sterile.
11. Females of childbearing potential who are taking contraceptive pills or agree to practice effective double barrier methods of contraception, from the time of signing the informed consent up to the last dose of study drug, and for 7 days after dosing stops, or who agree to completely abstain from heterosexual intercourse.
12. Capability of understanding, consenting to, and complying with study requirements, study visits, and to return to the clinic for follow-up evaluations as specified by the protocol.

Exclusion Criteria:

1. A history of unstable or inadequately treated medical illnesses including moderate to severe brain injury, or neurological illnesses impacting cognitive function. Patients with a personal or family history of cardiac problems will need to undergo EKG at screen visit, and will be excluded if results are abnormal.
2. Patients taking procognitive medications, clozapine, tricyclic antidepressants, first-generation antipsychotics, and cogentin.
3. Those taking two or more antipsychotics.
4. Those taking strong CYP3A4 inhibitors (e.g. clarithromycin, nefazodone, grapefruit juice) or strong CYP3A4 inducers (e.g. carbamazepine, St John's wort (Hypericum perforatum). Please refer to the current Lurasidone SmPC for further listed contraindications.
5. Anticholinergics and stimulants that increase dopamine levels are not permitted
6. Cognitive remediation therapy within 3 months prior to entry or during the double blind phase.
7. Neuromodulation treatment with ECT or rTMS or tDCS or DBS within eight weeks or treatment with an experimental drug within 30 days.
8. History of nonresponse or intolerance to lurasidone.
9. Psychotic disorder other than Bipolar Disorder.
10. Patients who currently meet criteria for anxiety disorder (GAD, OCD, Panic disorder, PTSD).
11. Those with a current or lifetime diagnosis of ADHD or other learning disorders.
12. Axis I diagnosis of alcohol/substance abuse or dependence within the past month.
13. Significant risk of harm to self or others.
14. Pregnancy or lactation.
15. Liver function tests (AST and ALT) three times the upper limit of normal.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in cognitive performance in Euthymic bipolar patients treated with Lurasidone vs Placebo adjunctive therapy. | 6 weeks
  Cognitive improvement will be measured by changes in composite cognitive score from baseline to endpoint, extracted from the International Society for Bipolar Disorders-Battery for Assessment of Neurocognition.

SECONDARY OUTCOMES:
Change in Depression | 6 weeks
  Montgomery Asberg Depression Rating Scale (MADRS) will be used to assess changes in bipolar depression from baseline to endpoint.
Change in Mania | 6 weeks
  The Young Mania Rating Scale (YMRS) will be used to assess changes in mania from baseline to endpoint.
Improvement in overall psychiatric status | 6 weeks
  Clinical Global Improvement Scale will be used to assess change from baseline to endpoint in overall psychiatric status.
Improvement in Quality of Life | 6 weeks
  Quality of Life, Bipolar Version Scale will be used to assess improvement in quality of life from baseline to endpoint.
Improvement in Subjective-rated Cognitive Functioning | 6 weeks
  Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA) will be used to assess changes in subjective cognitive functioning from baseline to endpoint.
Improvement in Objectively Rated Daily Functioning | 6 weeks
  Functioning Assessment Short Test (FAST) will be used to assess improvement in objectively rated daily functioning, defined as change in scores from baseline to endpoint.
Improvement in Subjectively Rated Daily Functioning | 6 weeks
  Sheehan Disability Scale (SDS) will be used to assess improvement in subjectively rated daily functioning, defined as change in scores from baseline to endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi N Yatham, MBBS,MRCPsy, Principal Investigator — University of British Columbia, Department of Psychiatry
Locations (9):
- United States (2):
  - The Brigham and Women's Hospital, Department of Psychiatry, Boston, Massachusetts
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- UBC Mood Disorders Center, Vancouver, British Columbia, Canada
- Japan (5):
  - Department of Psychiatry, University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Department of Neuropsychiatry, Kansai Medical University, Moriguchi-shi, Osaka
  - Department of Psychiatry, Hokkaido University Graduate School of Medicine, Kita-ku, Sapporo
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Department of Psychiatry, Fujita Health University School of Medicine, Aichi, Toyoake
- Institute of Psychiatry, Psychology and Neuroscience,King's College London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No